CLINICAL TRIAL: NCT02462122
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of IDP-118 in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP-118 in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-118A-302; NCT02615093 (obsolete NCT alias)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-118 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-118 Lotion
- IDP-118 Vehicle Lotion (Active Comparator): Vehicle Lotion
  Interventions: Drug: IDP-118 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-118 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-118 Lotion
Drug: IDP-118 Vehicle Lotion — Lotion
  Other Names: Vehicle
  Arms: IDP-118 Vehicle Lotion

SUMMARY:
Safety and Efficacy of IDP-118 in the treatment of plaque psoriasis

DETAILED DESCRIPTION:
A Phase 3, Multicenter, Double-Blind, Randomized, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of IDP-118 in the Treatment of Plaque Psoriasis

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a BSA of at least 3%, but no more than 12%. The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an IGA score of 3 or 4. (The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this assessment).

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, MD, Study Director — Valeant Pharmaceuticals
Locations (16):
- United States (16):
  - Valeant Site 5, Fremont, California
  - Valeant Site 2, Boynton Beach, Florida
  - Valeant Site 14, North Miami Beach, Florida
  - Valeant Site 13, Detroit, Michigan
  - Valeant Site 8, Warren, Michigan
  - Valeant Site 10, Fridley, Minnesota
  - Valeant Site 1, East Windsor, New Jersey
  - Valeant Site 4, Albuquerque, New Mexico
  - Valeant Site 12, New York, New York
  - Valeant Site 6, High Point, North Carolina
  - Valeant Site 3, Portland, Oregon
  - Valeant Site 7, Knoxville, Tennessee
  - Valeant Site 9, College Station, Texas
  - Valeant Site 15, Houston, Texas
  - Valeant Site 16, Houston, Texas
  - Valeant Site 11, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-118 Lotion | IDP-118 Vehicle Lotion
Started | 141 | 74
Completed | 120 | 61
Not Completed | 21 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-118 Lotion | IDP-118 Vehicle Lotion | Total
Number analyzed (Participants) | 141 | 74 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (14.84) | 51.8 (13.18) | 51.8 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 24 | 79
  Male | 86 | 50 | 136

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Treatment Success at Week 8
Description: Treatment success was defined as at least a 2-grade improvement from Baseline in IGA score and an IGA score equating to "Clear" or "Almost Clear". IGA was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | IDP-118 Vehicle Lotion
Number analyzed (Participants) | 141 | 74
percentage of participants | 45.33 | 12.51

2. Secondary Outcome: Percentage of Participants With Treatment Success at Weeks 12, 6, 4, and 2
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | IDP-118 Vehicle Lotion
Number analyzed (Participants) | 141 | 74
percentage of participants
  Week 12 | 33.35 | 8.84
  Week 6 | 37.53 | 8.24
  Week 4 | 26.96 | 1.36
  Week 2 | 9.77 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety analysis set included all participants who were randomized, received at least one confirmed dose of study drug, and had at least one post-baseline safety assessment.
Arm/Group | IDP-118 Lotion | IDP-118 Vehicle Lotion
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/73
Other Adverse Events (participants affected / at risk) | 13/137 | 4/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=137) | IDP-118 Vehicle Lotion (N=73)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 13 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.